CLINICAL TRIAL: NCT01015157
Title: Laparoscopic Roux-en-Y Gastric Bypass Outcomes With Systematic Gastric Stapling Line Reinforcement With Seamguard Biomaterial
Brief Title: Prospective Trial Using Gastric Stapling Line Reinforcement With Seamguard in Roux-en-Y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de l'Anjou (Other)
Responsible Party: Philippe Topart MD, Société de Chirurgie Viscérale, Clinique de l'Anjou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEAM1
Record Dates: First submitted 2009-08-05; First posted 2009-11-18 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Gastric Bypass
Keywords: Gastric bypass; staple line reinforcement; outcomes; per and postoperative blood loss
MeSH Terms: conditions — Progressive Encephalomyelitis with Rigidity; Postoperative Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard stapling without reinforcement (Active Comparator): Standard Echelon 60 linear stapling with GOLD cartridges
  Interventions: Procedure: Roux-en-Y laparoscopic gastric bypass for morbid obesity
- Seamguard gastric stapling line reinforcement (Active Comparator)
  Interventions: Procedure: Roux-en-Y laparoscopic gastric bypass for morbid obesity

INTERVENTIONS:
Procedure: Roux-en-Y laparoscopic gastric bypass for morbid obesity — Primary bariatric surgery. Standard laparoscopic procedure with linear stapling divising of the stomach (Echelon 60 stapler, GOLD cartridges) with or with Seamguard reinforcement
  Other Names: Gore Seamguard biomaterial staple line reinforcement

SUMMARY:
Study objectives :

Primary endpoint is to a assess the change in blood loss (originating from stapling the stomach) with the use of Seamguard reinforcement Secondary endpoint is to evaluate the difference in leak rate

Methods :

Prospective. Randomized study. Published data does not allow for clear determination of the number of patients required for the study. Based on our own experience. The investigators estimate that the average postoperative blood loss is 200ml with a standard deviation of 100ml over 3 days. Based on this assumption. A total number of patients (control + Seamguard groups) of 60 is required if the expected reduction of the mean drainage volume is 100ml and 82 patients for an expected drainage volume reduction of 85ml.

All patients candidates to a laparoscopic gastric bypass will be enrolled in the study Under the conditions this is a primary bariatric procedure (no revision allowed)., no history of hiatal surgery such as anti-reflux nor significant upper abdominal surgery. The only associated surgical procedure allowed is the cholecystectomy.

Patients' inclusion :

Will be done immediately before surgical procedure following acceptance of a written consent.

Bleeding from liver or slpeen injury will lead to patient's exclusion.

Methods :

Surgical procedures are identical for the 2 surgeons of the study (GB and PT) with 30-50ml gastric pouch. Linear. side to side. Antegastric and antecolic gastrojejunal anstomosis . Use of Echelon 60 linear stapler with GOLD cartridges on stomach. Blue to perform the gastrojejunal anastomosis and white on Small bowel. Peroperativeblood loss and need to apply clips or stitches on the gastric staple line are recorded. Operation time and patient information (BMI. Comorbidities) are recorded as well any noticeable or unexpected event.

Postoperative blood loss is assessed by at least 1 abdominal closed circuit suction drain left for a minimum of 3 days (removal on postop day 3 at the earliest).

In addition hemoglobin and red cell count is performed on postop day 1 and 2. Absence of leakage is confirmed by methylene blue test perop as well as on postop day 1 before resuming fluids and on postop day 2 by a gastrograffin swallow. Drinks and food are resumed according to the standard practice between postop day 1 and postop day 2.

Duration of the hospital stay and postoperative course will be documented. Early follow up is clinically done at 1 month postop without any specific radiological or biological examination.

Data collection Will be done on a form during and after the procedure

BLOOD LOSS : peroperative volume as well as daily drainage output (postop day 1. 2 and 3) as well as the sum of the 3 postop days.

Hemoglobin change is recorded on day 1 and 2. Need to leave drain(s) for more than 3 days is recorded.

Study completion :

Estimated time to complete the study based on the current experience is between 5 and 7 months. Sudy is closed 1 month after the last inclusion.

ELIGIBILITY:
Inclusion Criteria:

* all primary laparoscopic Roux-en-Y gastric bypasses for morbid obesity

Exclusion Criteria:

* additional procedures except cholecystectomy, peroperative bleeding from spleen or liver injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Blood loss volume per and postoperatively, additional hemostatic measures peroperatively, hemoglobin levels postoperatively | 3 days postoperatively

SECONDARY OUTCOMES:
gastrojejunal anastomosis leakage rate: clinical and radiological | postoperative day 2 (gastrograffin swallow)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Topart, MD, Principal Investigator — Société de Chirurgie Viscérale
Locations (1):
- Clinique de l'Anjou, Angers, France